CLINICAL TRIAL: NCT06401902
Title: Diabetes and Stroke: Does an Excess Risk of Hemodynamic Cerebral Ischemia Exist?
Brief Title: Diabetes and Risk of Ischemic Stroke.
Status: Completed | Type: Observational
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Other Study IDs: VASC-01-2024
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Carotid Stenosis
Keywords: diabetes; ischemic stroke; cerebral hemorrhage; hypoperfusion; hyperperfusion
MeSH Terms: conditions — Carotid Stenosis; Diabetes Mellitus; Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetics: Diabetics patients who underwent internal carotid artery surgery
  Interventions: Procedure: carotid clamping
- Nondiabetics: Nondiabetics patients who underwent internal carotid artery surgery
  Interventions: Procedure: carotid clamping

INTERVENTIONS:
Procedure: carotid clamping — Occurrence of consciousness perturbations, language difficulties and/or contralateral motor deficit during the carotid-clamping test and requiring shunt placement.

SUMMARY:
Diabetes in an independent risk factor for ischemic stroke, whose associated mortality rate is higher and sequelae more serious than for nondiabetics. Diabetes increases the risk of stroke or death after surgical carotid revascularization or endoluminal angioplasty. It is, with contralateral ICA occlusion, 1 of the 7 factors doubling the stroke risk after carotid endarterectomy. Diabetes also enhances the cerebral hemorrhage risk associated with carotid surgery, thrombectomy or thrombolysis revascularization of the cerebral arteries.

This study was undertaken to examine whether the hemodynamic cerebral ischemia (HCI) frequency, which increases stroke severity, is higher in diabetics than nondiabetics and, if diabetes carries an excess HCI risk, whether it is independent of contralateral ICA occlusion.

DETAILED DESCRIPTION:
Embolic and hemodynamic mechanisms are the main causes underlying ischemic strokes of carotid origin. The hemodynamic cerebral ischemia (HCI) risk depends on the contribution of the contralateral internal carotid artery (ICA) and vertebral arteries via the circle of Willis, the ipsilateral external carotid artery via the ophthalmic artery and the leptomeningeal arteries. During carotid surgery, impaired collateral flow is associated with the need for shunt insertion.

When HCI is present, cerebral perfusion is initially maintained by vasodilation of precapillary arterioles and the increased extraction coefficient of oxygen. Secondarily, vascular reserve exhaustion by degradation of arterial lesions engenders a loss of cerebral autoregulation, ischemic penumbra and cerebral infarction.

Carotid revascularization with an incomplete circle of Willis enhances the postoperative ischemic stroke risk. The loss of cerebral autoregulation, attributable to HCI combined with ipsilateral carotid tight stenosis, heightens the risk of hyperperfusion and cerebral hemorrhage.

Carotid occlusion is the primary cause of HCI. Carotid occlusions and tight stenoses lead to loss of cerebral autoregulation and cerebrovascular reserve, and have been associated with a 4-fold-increased stroke risk.

Diabetes in an independent risk factor for ischemic stroke, whose associated mortality rate is higher and sequelae more serious than for nondiabetics. Diabetes increases the risk of stroke or death after surgical carotid revascularization or endoluminal angioplasty.It is, with contralateral ICA occlusion, 1 of the 7 factors doubling the stroke risk after carotid endarterectomy. Diabetes also enhances the cerebral hemorrhage risk associated with carotid surgery, thrombectomy or thrombolysis revascularization of the cerebral arteries.

This study was undertaken to examine whether the HCI frequency is higher in diabetics than nondiabetics and, if diabetes carries an excess HCI risk, whether it is independent of contralateral ICA occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clamping test during carotid surgery.

Exclusion Criteria:

* Patients without clamping test during carotid surgery.

Ages: 28 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid stenosis requiring carotid surgery.
Sampling Method: Probability Sample
Enrollment: 3739 (Actual)
Dates: Start 1990-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Intolerance to carotid clamping test | During clamping test
  Occurrence of consciousness perturbations: patient loses consciousness
Intolerance to carotid clamping test. | During clamping test
  Language difficulties: the patient no longer answers questions
Intolerance to carotid clamping test. | During clamping test
  Contralateral motor deficit: anesthesiologist request to shake hands.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pr PETITJEAN, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Mutualist Montsouris Institute, Paris, Île-de-France Region, France